CLINICAL TRIAL: NCT03295279
Title: Pulmonary Diseases in WTC Workers: Symptoms, Function, and Chest CT Correlates
Brief Title: WTC Chest CT Imaging Archive
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of Pittsburgh (Other); Brigham and Women's Hospital (Other); National Jewish Health (Other)
Responsible Party: Principal Investigator, Rafael E. de la Hoz, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 12-0751; U01OH010401 (NIH); U01OH011697 (NIH); GCO 17-2598 (Other: Icahn School of Medicine at Mount Sinai); U01OH012782 (NIH); GCO 23-2259 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2017-09-25; First posted 2017-09-27 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Airway Disease; Interstitial Lung Disease; Lung Cancer
Keywords: World Trade Center; Quantitative computerized tomography; Qualitative computerized tomography of the chest; Chronic airway disease; Interstitial lung disease; Occupational pulmonology; Spirometry; Forced Oscillometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Dr. Rafael E de la Hoz and colleagues have performed standardized and computer-assisted readings of all chest CT scans received by WTC workers and volunteers at the Mount Sinai Medical Center between 2003 and 2016. The clinical team sought to assess all findings suggestive of airway, interstitial, and neoplastic disease in a systematic way, and correlate those findings with clinical, functional, and exposure indicators. The study team's research will also involve analyses of longitudinal imaging and functional trends, and characterization of the WTC related lower airway diseases and their risk factors, with a focus on obesity-related imaging markers. The study team also plans to characterize the transitions into chronic obstructive pulmonary disease (COPD) among these workers.

The researchers also propose to test the use of added respiratory surveillance tools and explore functional markers of disease progression, explore alternate methods to investigate longitudinal functional trajectories, and novel spirometry calibration methods that might facilitate the implementation of spirometry in nonspecialized settings.

DETAILED DESCRIPTION:
The goal of this proposal is to characterize WTC-related lower airway disorders, and use novel imaging approaches to the investigation of obesity, one of their most important risk factors for poor clinical outcome and chronicity. To that end, the clinical team will utilize the WTC Pulmonary Evaluation Unit Chest CT Imaging Archive, an already established large imaging database, linked to extensive related databases that include disease symptoms, both pre-WTC and WTC-related occupational exposures, detailed pulmonary function and longitudinal spirometry measurements, visual imaging classification and grading, and quantitative computer assisted method (QCAM) measurements of airway, pulmonary parenchymal, pleural, and cardiovascular abnormalities. During the course of the proposed research project, the clinical team will continue to enrich most sources of data with periodic updates, in order to accrue information on the trajectories of the different clinical, functional, and imaging abnormalities observed in this population, and investigate the role of key adverse risk factors directly, and in collaboration with other investigators. In a related project, the research team will focus on COPD, classifying its severity, investigating its diagnostic stability, progression, and transitions, characterize structural abnormalities as assessed by chest CT imaging, and examine the interaction of WTC-related exposure levels with tobacco smoking on increasing the risk of for the disease.

Grant U01 OH010401 was renewed to 6/30/2026.

Grant U01 OH011697 proposes (1) to establish the quantitative computed tomography (QCT) characteristics that may differentiate WTC-related from non-WTC-related COPD, (2) investigate characteristics and longitudinal lung function trajectories of WTC patients with pre-COPD, and (3) investigate lung mechanical strain (LMS) as an early QCT marker of lung injury associated with chronic disease and accelerated longitudinal lung function decline.

Grant U01 OH012782-01-00 proposes (1) to test the use of added respiratory surveillance tools (diffusion capacity and forced oscillometry) and explore functional markers of disease progression, (2) explore alternate methods to investigate longitudinal functional trajectories, and (3) novel spirometry calibration methods that might facilitate the implementation of spirometry in nonspecialized settings.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be participants in the screening/monitoring (SMP) and treatment program (TP) sides of the WTC Health Plan Clinical Center Excellence at Mount Sinai Medical Center, the major site, by far of the NY/NJ consortium of this program.

Exclusion Criteria:

* Special vulnerable populations, such as fetuses, neonates, pregnant women, children, prisoners, institutionalized individuals, will not be involved in this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will be participants in the screening/monitoring (SMP) and treatment program (TP) sides of the WTC Health Plan Clinical Center Excellence at Mount Sinai Medical Center, the major site, by far of the NY/NJ consortium of this program.
Sampling Method: Non-Probability Sample
Enrollment: 2122 (Estimated)
Dates: Start 2012-09-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Accelerated longitudinal FEV1 decline | 5 years
  The clinical team selects spirometries of acceptable quality, and subjects with at least 3 spirometries spanning at least 5 years, to calculate FEV1 slope, which can then be modeled quantitatively. For categorical analyses, the clinical team defines rapid FEV1 decliners and contrast them to normal-and-stable FEV1 subjects, defined as those having an FEV1 above the lower limit of normal at baseline, no bronchodilator response, and FEV1 not changing by more than 25 ml/year on average in either direction.

SECONDARY OUTCOMES:
Number of physician diagnosis of incident asthma | 5 years
  Physician diagnosis of asthma with onset after WTC occupational exposures.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael E. de la Hoz, MD, MPH, MSc, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Napier CO, Mbadugha O, Bienenfeld LA, Doucette JT, Lucchini R, Luna-Sanchez S, de la Hoz RE. Obesity and weight gain among former World Trade Center workers and volunteers. Arch Environ Occup Health. 2017 Mar 4;72(2):106-110. doi: 10.1080/19338244.2016.1197174. Epub 2016 Jun 7. PMID 27268046
- [Background] de la Hoz RE, Jeon Y, Miller GE, Wisnivesky JP, Celedon JC. Post-traumatic Stress Disorder, Bronchodilator Response, and Incident Asthma in World Trade Center Rescue and Recovery Workers. Am J Respir Crit Care Med. 2016 Dec 1;194(11):1383-1391. doi: 10.1164/rccm.201605-1067OC. PMID 27548615
- [Background] de la Hoz RE, Liu X, Doucette JT, Reeves AP, Bienenfeld LA, Wisnivesky JP, Celedon JC, Lynch DA, San Jose Estepar R. Increased Airway Wall Thickness is Associated with Adverse Longitudinal First-Second Forced Expiratory Volume Trajectories of Former World Trade Center workers. Lung. 2018 Aug;196(4):481-489. doi: 10.1007/s00408-018-0125-7. Epub 2018 May 24. PMID 29797069
- [Background] de la Hoz RE, Weber J, Xu D, Doucette JT, Liu X, Carson DA, Celedon JC. Chest CT scan findings in World Trade Center workers. Arch Environ Occup Health. 2019;74(5):263-270. doi: 10.1080/19338244.2018.1452712. Epub 2018 May 9. PMID 29543564
- [Background] de la Hoz RE, Jeon Y, Reeves AP, San Jose Estepar R, Liu X, Doucette JT, Celedon JC, Nolan A. Increased pulmonary artery diameter is associated with reduced FEV1 in former World Trade Center workers. Clin Respir J. 2019 Oct;13(10):614-623. doi: 10.1111/crj.13067. Epub 2019 Aug 19. PMID 31347281
- [Background] de la Hoz RE, Liu X, Celedon JC, Doucette JT, Jeon Y, Reeves AP, San Jose Estepar R. Association of Obesity with Quantitative Chest CT Measured Airway Wall Thickness in WTC Workers with Lower Airway Disease. Lung. 2019 Aug;197(4):517-522. doi: 10.1007/s00408-019-00246-z. Epub 2019 Jun 28. PMID 31254057
- [Background] de la Hoz RE. Occupational lower airway disease in relation to World Trade Center inhalation exposure. Curr Opin Allergy Clin Immunol. 2011 Apr;11(2):97-102. doi: 10.1097/ACI.0b013e3283449063. PMID 21325944
- [Background] de la Hoz RE, Shohet MR, Chasan R, Bienenfeld LA, Afilaka AA, Levin SM, Herbert R. Occupational toxicant inhalation injury: the World Trade Center (WTC) experience. Int Arch Occup Environ Health. 2008 Feb;81(4):479-85. doi: 10.1007/s00420-007-0240-x. Epub 2007 Sep 5. PMID 17786467
- [Background] Mendelson DS, Roggeveen M, Levin SM, Herbert R, de la Hoz RE. Air trapping detected on end-expiratory high-resolution computed tomography in symptomatic World Trade Center rescue and recovery workers. J Occup Environ Med. 2007 Aug;49(8):840-5. doi: 10.1097/JOM.0b013e3180d09e87. PMID 17693781
- [Background] Sigel KM, Xu D, Weber J, Wisnivesky JP, Celedon JC, de la Hoz RE. Prevalence of Pulmonary Nodules Detected by Computed Tomography in World Trade Center Rescue and Recovery Workers. Ann Am Thorac Soc. 2020 Jan;17(1):125-128. doi: 10.1513/AnnalsATS.201907-517RL. No abstract available. PMID 31499008
- [Background] Weber J, Reeves AP, Doucette JT, Jeon Y, Sood A, San Jose Estepar R, Celedon JC, de la Hoz RE. Quantitative CT Evidence of Airway Inflammation in WTC Workers and Volunteers with Low FVC Spirometric Pattern. Lung. 2020 Jun;198(3):555-563. doi: 10.1007/s00408-020-00350-5. Epub 2020 Apr 1. PMID 32239319
- [Background] de la Hoz RE, Shapiro M, Nolan A, Celedon JC, Szeinuk J, Lucchini RG. Association of low FVC spirometric pattern with WTC occupational exposures. Respir Med. 2020 Aug-Sep;170:106058. doi: 10.1016/j.rmed.2020.106058. Epub 2020 Jun 7. PMID 32843177
- [Derived] Sigel K, de la Hoz RE, Markowitz SB, Kong CY, Stone K, Todd AC, Wisnivesky JP. Lung cancer incidence among world trade center rescue and recovery workers. Cancer Med. 2022 Aug;11(16):3136-3144. doi: 10.1002/cam4.4672. Epub 2022 Mar 28. PMID 35343066
- See also: Principal investigator's ORCID record — http://orcid.org/0000-0002-8949-9279/print
- See also: Principal investigator's WTC-related bibliography — https://www.ncbi.nlm.nih.gov/sites/myncbi/1t5YX2bFtgN/collections/58762945/public/
- See also: Principal investigator's RePORT site for Study 24-00850 — https://reporter.nih.gov/search/MY8RCxAMMU2ClUwp6cBY4Q/project-details/10995057
- See also: Principal investigator's RePORT site for Study 12-00925 — https://reporter.nih.gov/search/MY8RCxAMMU2ClUwp6cBY4Q/project-details/10848174
- See also: Principal investigator's RePORT site for Study 18-00595 — https://reporter.nih.gov/search/MY8RCxAMMU2ClUwp6cBY4Q/project-details/10886482